CLINICAL TRIAL: NCT01553721
Title: A Placebo-controlled, Double-blind, Phase II Clinical Study to Evaluate the Efficacy and Safety of Udenafil in Patient With Pulmonary Arterial Hypertension(PAH)
Brief Title: Efficacy and Safety Study of Udenafil in Patient With Pulmonary Arterial Hypertension(PAH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DA8159_PAH_II
Record Dates: First submitted 2012-01-01; First posted 2012-03-14 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — udenafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- udenafil (Experimental): 1. Phase IIa Experimental : Udenafil Dose 1, Dose 2
  2. Phase IIb Experimental : Udenafil
  Interventions: Drug: udenafil
- placebo (Placebo Comparator): 1. Phase IIa Placebo Comparator : Placebo
  2. Phase IIb Placebo Comparator : Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: udenafil — Phase IIa - Udenafil Dose 1, Dose 2(Single dose)
  Phase IIb - Udenafil(BID)
  Arms: udenafil
Drug: placebo — Phase IIa - placebo Phase IIb - placebo
  Arms: placebo

SUMMARY:
This is a placebo-controlled, double-blind, phase II clinical study to evaluate the efficacy and safety of Udenafil in patient with Pulmonary Arterial Hypertension(PAH).

ELIGIBILITY:
Inclusion Criteria:

• Subjects aged 18 and over who have any of the following diseases

* primary Pulmonary Arterial Hypertension
* secondary Pulmonary Arterial Hypertension caused by connective tissue disease
* [Phase IIb] Pulmonary Arterial Hypertension caused by congenital heart disease(including Eisenmenger syndrome)

Exclusion Criteria:

* Subjects with pulmonary arterial hypertension caused by any etiology other than those specified in the inclusion criteria
* BMI(Body Mass Index) < 18.5kg/m2
* Subjects with hypotension(SBP/DBP<90/50mmHg) or uncontrolled hypertension(SBP/DBP>170/100mmHg)
* Creatinine clearance ≤ 30mL/min
* History of non-arteritic anterior ischemic optic neuropathy(NAION)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2011-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Phase IIa - Pulmonary vascular resistance index(PVRI) | 4 hours
Phase IIb - 6-minute walk distance | 16weeks

CONTACTS AND LOCATIONS:
Overall Officials: Duk-Kyung Kim, M.D., Ph.D, Principal Investigator — Samsung Medical Center, 50 Irwon-Dong, Gangnam-Gu, Special city of Seoul, 135-710, Korea
Locations (9):
- South Korea (9):
  - Seoul National University Hospital, Seoul, Chongno-gu, 28 Yongon-dong
  - Samsung Medical Center, Seoul, Gangnam-Gu, Irwon-Dong 50
  - Severance Hospital, Yonsei University Health System, Special City of Seoul, Seodaemungu, 250 Seonsanno
  - Chungbook national University Hospital, Chungju
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Pusan national University Hospital, Pusan
  - Asan Medical Center, Seoul
  - The catholic univ. of korea Seoul ST. MARY's hospital, Seoul

REFERENCES:
- [Derived] Chang HJ, Song S, Chang SA, Kim HK, Jung HO, Choi JH, Lee JS, Kim KH, Jeong JO, Lee JH, Kim DK. Efficacy and Safety of Udenafil for the Treatment of Pulmonary Arterial Hypertension: a Placebo-controlled, Double-blind, Phase IIb Clinical Trial. Clin Ther. 2019 Aug;41(8):1499-1507. doi: 10.1016/j.clinthera.2019.05.006. Epub 2019 Jun 13. PMID 31202506
- [Derived] Chang SA, Kim HK, Chang HJ, Kim DK. Acute Hemodynamic Changes after Single Administration of Udenafil in Pulmonary Arterial Hypertension: a Phase IIa Study. Korean Circ J. 2019 Apr;49(4):353-360. doi: 10.4070/kcj.2018.0281. Epub 2018 Dec 10. PMID 30808080